CLINICAL TRIAL: NCT07314476
Title: CardioLogical Interventions and Acute strOke Treatment sTudy
Acronym: CLOT
Status: Not yet recruiting | Type: Observational
Sponsor: University of L'Aquila (Other)
Collaborators: Rete delle NeuroCardiologie (Unknown)
Responsible Party: Principal Investigator, Simona Sacco, Full Professor of Neurology, University of L'Aquila
Other Study IDs: 1.0 - 08/02/2025
Record Dates: First submitted 2025-12-02; First posted 2026-01-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke AIS; Stroke Treatment; PCI Patients; Aortic Valve Replacement; Transcatheter Aortic Valve Replacement (TAVR); Mitral Valve Repair; Mitral Valve Replacement; Left Atrial Appendage Closure; Transcatheter Pulmonary Valve Replacement (TPVR)
Keywords: acute ischemic stroke; acute ischemic stroke treatments; cardiological intervention
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 180 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with ischemic stroke occuring within 28 days after cardiological interventional procedures: Cardiological interventions includes: Percutaneuous Coronary Intervention - PCI, Transcatheter Aortic Valve Replacement - TAVR, Baloon Aortic Valvuloplasy - BAV, Percutaneous Mitral Valve Repair or Replacement, Patent Formaen Ovale - PFO - or Atrial Septal Defects - ASD - Closure, Left Atrial Appendage Closure, Transcatheter Pulmonary Valve Replacement, Percutaneous Closure of Paravalvular Leaks

SUMMARY:
The study aims to investigate characteristics and prognosis of ischemic stroke cases following cardiological interventions, focusing on the effectiveness and safety of acute ischemic stroke treatments.

DETAILED DESCRIPTION:
CLOT is a multicenter, observational, ambispective real-world study involving acute ischemic stroke cases occuring after cardiological procedures.

Patients will be recruited at different emergency services and stroke units in Europe. The study will encompass a retrospective (CLOT-R) and prospective (CLOT-P) data collection.

CLOT-R will include cases the occured in the 5 years befor the initation of the study; CLOT-P has a duration of 2 years of enrollement from the study approval at each site and follow-up of 180 days (total duration of 2 years and 180 days). The inclusion criteria are: acute ischemic stroke in adult patient (18 years of age or older) as diagnosed according to the World Health Organization (WHO) criteria; stroke with evidence of CT/MRI DWI/FLAIR acute lesion in the first neuroimaging or in the follow-up at 24-48 h; interventional cardiological procedures performed within 28 days since the stroke onset (Percutaneuous Coronary Intervention - PCI, Transcatheter Aortic Valve Replacement - TAVR, Baloon Aortic Valvuloplasy - BAV, Percutaneous Mitral Valve Repair or Replacement, Patent Formaen Ovale - PFO - or Atrial Septal Defects - ASD - Closure, Left Atrial Appendage Closure, Transcatheter Pulmonary Valve Replacement, Percutaneous Closure of Paravalvular Leaks); written informed consent provided by the patient himself or by proxy (for unconscious patients, cognitively impaired, or aphasic).

Exclusion criteria are: Stroke-like symptoms due primarily to another non-ischemic/hemorrhagic acute neurological condition or stroke mimics (e.g. severe hypo- or hyperglycemia, migraine with aura, functional disorders, etc); Spontaneous and post traumatic hemorrhagic stroke or spontaneous/post-traumatic subarachnoid hemorrhage or subdural hematoma; Impossibility to achieve written informed consent.

The primary outcome of CLOT-R is a descriptive analysis of baseline demographic, clinical, neuroimaging, cardiological procedural and acute stroke treatment characteristics. The secondary outcomes are: effectiveness and safety of intravenous thrombolysis (IVT) with or without mechanical thrombectomy (MT), or MT alone; 90-day post-stroke risk of all-cause and vascular mortality, new ischemic stroke or transient ischemic attack (TIA), myocardial infarction, intracranial hemorrhage or other major bleeding events, disability as measured by the modified Rankin Scale (mRS) score.

The primary outcome of CLOT-P is effectiveness and safety of IVT with or without MT, or MT alone. The secondary outcomes are 90-day and 180-day post-stroke risk of all-cause and vascular mortality, new ischemic stroke or TIA, myocardial infarction, intracranial hemorrhage or other major bleeding events, disability as measured by the mRS score.

The statistic analyses will include Descriptive statistics (baseline characteristics), Poisson regression analysis (incidence of primary and secondary outcomes at each timepoint), Cox regression analysis (time-to-outcomes comparison between groups, identification of outcomes predictors), generalized linear regression (ordinal mRS distribution comparison between maintainers and switchers), risk ratio and risk difference calculation for primary and secondary outcomes comparison (unadjusted and adjusted for confounders), pseudo-randomization (propensity score matching or inverse probability weighting).

The study aims to include in CLOT-P a minimum sample of 400 patients (100 patients for each acute stroke treatment group and 100 untreated) to have reliable estimates of the primary study outcome.

ELIGIBILITY:
Inclusion Criteria:

* acute ischemic stroke in adult patient (18 years of age or older) as diagnosed according to the World Health Organization (WHO) criteria;
* stroke with evidence of CT/MRI DWI/FLAIR acute lesion in the first neuroimaging or in the follow-up at 24-48 h;
* interventional cardiological procedures performed within 28 days since the stroke onset (Percutaneuous Coronary Intervention - PCI, Transcatheter Aortic Valve Replacement - TAVR, Baloon Aortic Valvuloplasy - BAV, Percutaneous Mitral Valve Repair or Replacement, Patent Formaen Ovale - PFO - or Atrial Septal Defects - ASD - Closure, Left Atrial Appendage Closure, Transcatheter Pulmonary Valve Replacement, Percutaneous Closure of Paravalvular Leaks);
* written informed consent provided by the patient himself or by proxy (for unconscious patients, cognitively impaired, or aphasic).

Exclusion Criteria:

* Stroke-like symptoms due primarily to another non-ischemic/hemorrhagic acute neurological condition or stroke mimics (e.g. severe hypo- or hyperglycemia, migraine with aura, functional disorders, etc);
* Spontaneous and post traumatic hemorrhagic stroke or spontaneous/post-traumatic subarachnoid hemorrhage or subdural hematoma;
* AciuImpossibility to achieve written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke in adult patient (>18 years old) after cardiological intervention, male and female.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
CLOT-R primary outcome - Stroke severity | from enrollment to 180 days follow-up
  Stroke severity assessed via the National Institutes of Health Stroke Scale (NIHSS). Scores on the NIHSS range from 0 to 42, with higher scores indicating more severe neurological deficits.
CLOT-R primary outcome - Radiology | from enrollment to 180-day follow-up
  Number of participants with large vessel occlusion demonstrated on neuroimaging.
CLOT-R primary outcome - Cardiological procedure | from enrollment to 180-day follow-up
  Number of participants who underwent cardiological procedures during which ischemic stroke occurred.
CLOT-P primary outcome - Efficacy | 90-day follow-up
  Number of participants presenting with Modified Rankin Scale (mRS) score ≤2 after revascularization. Scores on the mRS range from 0 to 6, with 0 indicating no symptoms and 6 indicating death. A score of 2 or less indicates functional indipendence.
CLOT-P primary outcome - safety | 90-day follow-up
  Number of participants with symptomatic intracranial hemorrhage after revascularization.

SECONDARY OUTCOMES:
CLOT-R secondary outcome - Efficacy | 90-day follow-up
  Number of participants presenting with Modified Rankin Scale (mRS) score ≤2 after revascularization. Scores on the mRS range from 0 to 6, with 0 indicating no symptoms and 6 indicating death. A score of 2 or less indicates functional indipendence.
CLOT-R secondary outcome - Safety | 90-day follow-up
  Number of patients with symptomatic intracranial hemorrhage after revascularization.
CLOT-R secondary outcome: Serious Adverse Event (SAE) | 90-day follow-up
  Number of patients experiencing Serious Adverse Events (retrospective investigation).
CLOT-P secondary outcome: Serious Adverse Event (SAE) | 90-day and 180-day follow-up
  Number of patients experiencing Serious Adverse Events (prospective investigation).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Biotechnological and Applied Clinical Sciences, L’Aquila, L'Aquila, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] D'Anna L, Demir O, Banerjee S, Malik I. Intravenous Thrombolysis and Mechanical Thrombectomy in Patients with Stroke after TAVI: A Report of Two Cases. J Stroke Cerebrovasc Dis. 2019 Oct;28(10):104277. doi: 10.1016/j.jstrokecerebrovasdis.2019.06.035. Epub 2019 Jul 18. PMID 31327683
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL. Guidelines for the Early Management of Patients With Acute Ischemic Stroke: 2019 Update to the 2018 Guidelines for the Early Management of Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2019 Dec;50(12):e344-e418. doi: 10.1161/STR.0000000000000211. Epub 2019 Oct 30. PMID 31662037
- [Background] Shah R, Wilkins E, Nichols M, Kelly P, El-Sadi F, Wright FL, Townsend N. Epidemiology report: trends in sex-specific cerebrovascular disease mortality in Europe based on WHO mortality data. Eur Heart J. 2019 Mar 1;40(9):755-764. doi: 10.1093/eurheartj/ehy378. PMID 30124820
- [Background] D'Anna L, Abu-Rumeileh S, Merlino G, Ornello R, Foschi M, Diana F, Barba L, Mastrangelo V, Romoli M, Lobotesis K, Bax F, Kuris F, Valente M, Otto M, Korompoki E, Sacco S, Gigli GL, Nguyen TN, Banerjee S. Safety and Outcomes of Mechanical Thrombectomy in Acute Ischemic Stroke Attributable to Cardiological Diseases: A Scoping Review. J Am Heart Assoc. 2024 Sep 3;13(17):e034783. doi: 10.1161/JAHA.124.034783. Epub 2024 Jun 14. PMID 38874062